CLINICAL TRIAL: NCT03360669
Title: Comparison of Blood Pressure Measurement With an Omron HEM-907 Device in a Clinical Setting and a Research Setting
Acronym: OMRONHEM-907
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Maxime Lamarre-Cliche, MD, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: OMRON HEM-907
Record Dates: First submitted 2017-11-17; First posted 2017-12-04 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Hypertension
Keywords: hypertension, blood pressure, systolic, diastolic, AOBP, Omron HEM-907, research, clinical
MeSH Terms: conditions — Hypertension; Systolic Murmurs; Heart Murmurs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence: Clinical/Research (Experimental): Participants assigned to this arm will have their blood pressure measured in a clinical setting first, and in a research setting second. The sequence randomization corresponds to the intervention. Visits will be at least a day apart but within a two-week period. During the clinical visit, they will have their blood pressure measured with the Omron HEM-907, an automated office blood pressure (AOBP) device. During the research setting, participants will be guided through a series of research-driven steps such as study questionnaires and completion of consent forms. They will have their blood pressure measured in both arms with a mercury sphygmomanometer, and then 3 measurements with a mercury sphygmomanometer. AOBP measurements (Omron HEM-907) will be performed at the end of the visit.
  Interventions: Other: Sequence: Clinical/Research
- Sequence: Research/Clinical (Active Comparator): Participants assigned to this arm will go through the same measurements and procedures exception made of the research-first and clinical-second sequence. The intervention to which they are randomized corresponds to the sequence of the visits.
  Interventions: Other: Sequence: Research/Clinical

INTERVENTIONS:
Other: Sequence: Clinical/Research — Participants will be assigned to a sequence of: research visit first/clinical visit second.
  Arms: Sequence: Clinical/Research
Other: Sequence: Research/Clinical — Participants will be assigned to a sequence of: clinical visit first/research visit second.
  Arms: Sequence: Research/Clinical

SUMMARY:
Automated office blood pressure (AOBP) devices are recommended for high blood pressure diagnosis. One of those devices is the Omron HEM-907 (Omron Healthcare). It is currently not known if blood pressure measurements performed with this device in a clinical setting are equivalent to those made in a research setting. Therefore, this randomized-controlled trial was designed. It aims to compare the blood pressure measurements performed in a clinical and a research setting. Seventy patients will be included and randomized to a clinical/research or research/clinical sequence.

DETAILED DESCRIPTION:
Hypertension is a common condition, with an estimated prevalence around 20 percent in Canada. It is a major risk factor for cardiovascular disease. Recently, Hypertension Canada has updated its guidelines and recommend we should consider a 120 mm Hg systolic blood pressure target in high-risk patients aged 50 years or older. This recommendation derives mainly from the SPRINT trial. In this trial, blood pressure was measured with an automated oscillometric blood pressure (AOBP) device, the Omron HEM-907 (Omron Healthcare). However, it is not known if measurements performed with this device in a clinical setting are equivalent to those made in a research setting. Therefore, this randomized-controlled trial was designed. It aims to compare the blood pressure measurements of 70 patients in a clinical and a research setting. Patients will be randomized to a clinical/research or a research/clinical sequence.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Hypertensive or presumed hypertensive
* Patients with a scheduled visit at the IRCM hypertension clinic.

Exclusion Criteria:

* Limitation preventing the measurement of blood pressure
* Introduction or withdrawal of any blood pressure-modifying medication starting 4 weeks before the first and until the last study visit.
* Recreative drug use (except cannabis)
* Alcohol use of more than 4 drinks during the day
* New symptoms during the research visit, that warrants a medical evaluation
* Mean systolic blood pressure >180 mm Hg or mean diastolic blood pressure >110 mm Hg (using AOBP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Mean automated office blood pressure systolic blood pressure estimates | Up to 2 weeks

SECONDARY OUTCOMES:
Mean automated office blood pressure diastolic blood pressure estimates. | Up to 2 weeks
Individual unaveraged automated office systolic and diastolic blood pressure measurements (1, 2 and 3) | Up to 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Institut de Recherches Cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
according to specific scientifically pertinent demands

REFERENCES:
- [Background] Padwal RS, Bienek A, McAlister FA, Campbell NR; Outcomes Research Task Force of the Canadian Hypertension Education Program. Epidemiology of Hypertension in Canada: An Update. Can J Cardiol. 2016 May;32(5):687-94. doi: 10.1016/j.cjca.2015.07.734. Epub 2015 Aug 15. PMID 26711315
- [Background] Kannel WB. Blood pressure as a cardiovascular risk factor: prevention and treatment. JAMA. 1996 May 22-29;275(20):1571-6. PMID 8622248
- [Background] Ettehad D, Emdin CA, Kiran A, Anderson SG, Callender T, Emberson J, Chalmers J, Rodgers A, Rahimi K. Blood pressure lowering for prevention of cardiovascular disease and death: a systematic review and meta-analysis. Lancet. 2016 Mar 5;387(10022):957-967. doi: 10.1016/S0140-6736(15)01225-8. Epub 2015 Dec 24. PMID 26724178
- [Background] Pickering TG, James GD, Boddie C, Harshfield GA, Blank S, Laragh JH. How common is white coat hypertension? JAMA. 1988 Jan 8;259(2):225-8. PMID 3336140
- [Background] Myers MG, Valdivieso MA. Use of an automated blood pressure recording device, the BpTRU, to reduce the "white coat effect" in routine practice. Am J Hypertens. 2003 Jun;16(6):494-7. doi: 10.1016/s0895-7061(03)00058-x. PMID 12799100
- [Background] Edwards C, Hiremath S, Gupta A, McCormick BB, Ruzicka M. BpTRUth: do automated blood pressure monitors outperform mercury? J Am Soc Hypertens. 2013 Nov-Dec;7(6):448-53. doi: 10.1016/j.jash.2013.07.002. Epub 2013 Aug 19. PMID 23969286
- [Background] Leung AA, Daskalopoulou SS, Dasgupta K, McBrien K, Butalia S, Zarnke KB, Nerenberg K, Harris KC, Nakhla M, Cloutier L, Gelfer M, Lamarre-Cliche M, Milot A, Bolli P, Tremblay G, McLean D, Tran KC, Tobe SW, Ruzicka M, Burns KD, Vallee M, Prasad GVR, Gryn SE, Feldman RD, Selby P, Pipe A, Schiffrin EL, McFarlane PA, Oh P, Hegele RA, Khara M, Wilson TW, Penner SB, Burgess E, Sivapalan P, Herman RJ, Bacon SL, Rabkin SW, Gilbert RE, Campbell TS, Grover S, Honos G, Lindsay P, Hill MD, Coutts SB, Gubitz G, Campbell NRC, Moe GW, Howlett JG, Boulanger JM, Prebtani A, Kline G, Leiter LA, Jones C, Cote AM, Woo V, Kaczorowski J, Trudeau L, Tsuyuki RT, Hiremath S, Drouin D, Lavoie KL, Hamet P, Gregoire JC, Lewanczuk R, Dresser GK, Sharma M, Reid D, Lear SA, Moullec G, Gupta M, Magee LA, Logan AG, Dionne J, Fournier A, Benoit G, Feber J, Poirier L, Padwal RS, Rabi DM; Hypertension Canada. Hypertension Canada's 2017 Guidelines for Diagnosis, Risk Assessment, Prevention, and Treatment of Hypertension in Adults. Can J Cardiol. 2017 May;33(5):557-576. doi: 10.1016/j.cjca.2017.03.005. Epub 2017 Mar 10. PMID 28449828
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Myers MG, Godwin M, Dawes M, Kiss A, Tobe SW, Grant FC, Kaczorowski J. Conventional versus automated measurement of blood pressure in primary care patients with systolic hypertension: randomised parallel design controlled trial. BMJ. 2011 Feb 7;342:d286. doi: 10.1136/bmj.d286. PMID 21300709
- [Background] Myers MG, Oh PI, Reeves RA, Joyner CD. Prevalence of white coat effect in treated hypertensive patients in the community. Am J Hypertens. 1995 Jun;8(6):591-7. doi: 10.1016/0895-7061(95)00049-U. PMID 7662244
- [Background] Myers MG, Valdivieso M, Kiss A. Consistent relationship between automated office blood pressure recorded in different settings. Blood Press Monit. 2009 Jun;14(3):108-11. doi: 10.1097/MBP.0b013e32832c5167. PMID 19417634
- [Background] Agarwal R. Implications of Blood Pressure Measurement Technique for Implementation of Systolic Blood Pressure Intervention Trial (SPRINT). J Am Heart Assoc. 2017 Feb 3;6(2):e004536. doi: 10.1161/JAHA.116.004536. PMID 28159816